CLINICAL TRIAL: NCT04993950
Title: Effects of Sustained Natural Apophyseal Glides Along With Thoracic Postural Correction Techniques in Patients With Chronic Cervicogenic Headache
Brief Title: Effects of SNAGS Along With Thoracic Postural Correction Techniques in Patients With Chronic Cervicogenic Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/01008 Urooj Sajjad
Record Dates: First submitted 2021-08-05; First posted 2021-08-06 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Cervicogenic Headache
Keywords: cervicogenic headache, thoracic posture correction, SNAGS
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sustained natural apophyseal glides (Experimental): SNAGS will be applied in flexion, extension and rotation for a few seconds with 3 repetitions on the first day and 10 repetitions from the next visit.
  Interventions: Other: sustained natural apophyseal glides; Other: SNAGS with thoracic postural correction techniques
- SNAGS with thoracic postural correction techniques (Active Comparator): active as well as therapist-facilitated stretches.thoracic extension in sitting, Wall angle stretch and Corner stretch, while the therapist-facilitated stretches will be seated mid-thoracic stretch and prone mid thoracic stretch. Stretches will be maintained for 15-20 seconds with 10 repetitions of each stretch per session
  Interventions: Other: sustained natural apophyseal glides; Other: SNAGS with thoracic postural correction techniques

INTERVENTIONS:
Other: sustained natural apophyseal glides — SNAGS will be applied in flexion, extension and rotation for a few seconds with 3 repetitions on the first day and 10 repetitions from the next visit.
Other: SNAGS with thoracic postural correction techniques — thoracic extension in sitting, Wall angle stretch and Corner stretch, while the therapist-facilitated stretches will be seated mid-thoracic stretch and prone mid thoracic stretch. Stretches will be maintained for 15-20 seconds with 10 repetitions of each stretch per session

SUMMARY:
The aim of this study is to find out the effects of Mulligan SNAGs along with thoracic postural correction techniques on patients with chronic cervicogenic headache. Patients suffering from cervicogenic headache are often associated with muscle imbalance. This study will be significant in determining the effects of SNAGs along with thoracic postural correction techniques to improve pain, level of disability and functional status in patients of cervicogenic headache.

It will be Randomized controlled trial study design Data will be collected from Lady reading Hospital Peshawar Purposive sampling, group randomization using lottery method will be used in this study.

DETAILED DESCRIPTION:
Headaches are a common condition affecting 47% of the global population,1,2 with cervicogenic headaches (CGHs) accounting for 15-20% of all chronic and recurrent headaches. The International Headache Society has classified a cervicogenic headaches as a secondary headache with 'pain referred from a source in the neck and perceived in one or more regions of the head and/or face. In the case of cervicogenic headache, the cause is a disorder of the cervical spine and its component bone, disc and/or soft tissue elements. The term cervicogenic headache is commonly misused and does not simply apply to a headache associated with neck pain; many headache disorders, including migraine and tension-type headache, can have associated neck pain/tension. Rather, there must be evidence of a disorder or lesion within the cervical spine or soft tissues of the neck, known to be able to cause a headache (1). It is often worsened by neck movement, sustained awkward head position or external pressure over the upper cervical or occipital region the symptomatic side (2). The prevalence of Chronic headache has been reported to be between 0.4 and 20 % of the headache population (3). In recent years, there has been an increasing knowledge in the pathogenesis and better management of chronic headaches.

Current scientific evidence supports the role of manual therapies in the management of tension type and cervicogenic headache (4). Individuals with Chronic headache are frequently treated with spinal manipulative therapy including both mobilization and manipulation. Spinal mobilization consists of slow, rhythmical, oscillating techniques (5) Cervical sustained natural apophyseal glides (SNAGs) are 'mobilization with movement' technique in which a sustained accessory facet glide is applied together with active physiological movement. The therapist may apply the glide over the spinous process (central SNAGs) or over the articular pillar on one side (unilateral SNAGs). SNAGs have been advocated for the treatment of neck pain and range of movement (ROM) restriction. SNAGs have been shown to be effective for the treatment of neck pain, cervicogenic headaches, and cervicogenic dizziness (6).mobilization with movement utilize the dual role of bot therapist force (accessory glides) and patient effort (active physiological or functional movement) and techniques are often carried out in a variety of weight bearing positions, with treatment belts, and either additional therapist, assistant or patient applied overpressure A thorough clinical examination is performed and appropriate level is identified, the glide is then performed parallel to the perceived facet plane and the degree of glide is determined by patient's active movement response (8). Many studies on the short-term effectiveness and manual therapy to the cervical spine (mobilization and manipulative therapy) have found it beneficial in reducing headache pain or disability, intensity, frequency, and duration.

ELIGIBILITY:
Inclusion Criteria:

* Patients having headache for the last three months
* Patients having unilateral neck pain along with stiffness.
* A headache that is more frequent periorbitally, spreading to the temporal and ocular region and in the low occipital and less frequent in the frontal, parietal and facial region.
* Pain that is usually elicited by applying external pressure on at least 1 of the upper cervical joints (C0-C3) and moderate to severe non throbbing pain

Exclusion Criteria:

* Other types of headaches
* Congenital conditions of the cervical spine
* Disc herniation
* Cervical Fractures
* Degenerating disease of the cervical spine.
* Patients with contraindications to mobilization techniques and those with dizziness due to vertebrobasilar insufficiency or vestibular dysfunctions

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 38 (Actual)
Dates: Start 2022-02-20 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-20 (Actual)

PRIMARY OUTCOMES:
Visual Analog scale (VAS) | four weeks
  The VAS is a 10- cm graduated line. Each participant will self-assess the intensity of her pain. Patients in each group will be instructed to point to the position on the line between the faces to indicate how much pain they are currently feeling. The far-left end indicates "no pain" and the far right end indicates worst pain ever
Neck Disability Index (NDI) | for four weeks
  The NDI can be scored as a raw score or doubled and expressed as a percent. Each section is scored on a 0 to 5 rating scale, in which zero means 'No pain' and 5 means 'Worst imaginable pain.
Headache Impact Test | for four weeks
  Headache Impact Test is a tool used to measure the impact headaches have on your ability to function on the job, at school, at home and in social situations. Your score shows you the effect that headaches have on normal daily life and your ability to function.
Cervical ROM --Universal Goniometer | four weeks
  A large universal goniometer having a stationary arm and a moving arm of 12 inch and full circle body will be used for measuring cervical range of motion.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Khalid, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Lady reading Hospital, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Racicki S, Gerwin S, Diclaudio S, Reinmann S, Donaldson M. Conservative physical therapy management for the treatment of cervicogenic headache: a systematic review. J Man Manip Ther. 2013 May;21(2):113-24. doi: 10.1179/2042618612Y.0000000025. PMID 24421621
- [Background] Chaibi A, Russell MB. Manual therapies for cervicogenic headache: a systematic review. J Headache Pain. 2012 Jul;13(5):351-9. doi: 10.1007/s10194-012-0436-7. Epub 2012 Mar 30. PMID 22460941
- [Background] Dunning JR, Butts R, Mourad F, Young I, Fernandez-de-Las Penas C, Hagins M, Stanislawski T, Donley J, Buck D, Hooks TR, Cleland JA. Upper cervical and upper thoracic manipulation versus mobilization and exercise in patients with cervicogenic headache: a multi-center randomized clinical trial. BMC Musculoskelet Disord. 2016 Feb 6;17:64. doi: 10.1186/s12891-016-0912-3. PMID 26852024
- [Background] Fernandez-de-Las-Penas C, Courtney CA. Clinical reasoning for manual therapy management of tension type and cervicogenic headache. J Man Manip Ther. 2014 Feb;22(1):44-50. doi: 10.1179/2042618613Y.0000000050. PMID 24976747
- [Background] McDowell JM, Johnson GM, Hetherington BH. Mulligan Concept manual therapy: standardizing annotation. Man Ther. 2014 Oct;19(5):499-503. doi: 10.1016/j.math.2013.12.006. Epub 2014 Jan 10. PMID 24491791
- [Background] McDonnell MK, Sahrmann SA, Van Dillen L. A specific exercise program and modification of postural alignment for treatment of cervicogenic headache: a case report. J Orthop Sports Phys Ther. 2005 Jan;35(1):3-15. doi: 10.2519/jospt.2005.35.1.3. PMID 15754599
- [Background] Tul Ain SQ, Shakil Ur Rehman S, Maryam M, Kiani SK. Effects of Sustained Natural Apophyseal Glides with and without thoracic posture correction techniques on mechanical back pain: a randomized control trial. J Pak Med Assoc. 2019 Nov;69(11):1584-1587. doi: 10.5455/JPMA.274875.. PMID 31740859
- [Background] Reid SA, Callister R, Katekar MG, Rivett DA. Effects of cervical spine manual therapy on range of motion, head repositioning, and balance in participants with cervicogenic dizziness: a randomized controlled trial. Arch Phys Med Rehabil. 2014 Sep;95(9):1603-12. doi: 10.1016/j.apmr.2014.04.009. Epub 2014 May 2. PMID 24792139
- [Background] Vernon H. The Neck Disability Index: state-of-the-art, 1991-2008. J Manipulative Physiol Ther. 2008 Sep;31(7):491-502. doi: 10.1016/j.jmpt.2008.08.006. PMID 18803999